CLINICAL TRIAL: NCT05239689
Title: Clinical Study on the Safety and Effectiveness of CD38 CAR-T Cells in the Treatment of CD38-positive Hematological Malignancies
Brief Title: Clinical Study of CD38 CAR-T Cells in the Treatment of Hematological Malignancies
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, The President of The First Affiliated Hospital, College of Medicine, Zhejiang University, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD38-001
Record Dates: First submitted 2021-12-01; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: AML
Keywords: AML; CD38 CAR T-cell therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment of CD38-positive Hematological Malignancies (Experimental): Administration of CD38 CAR T-cells A dose levels of 2-8*10E6/kg are administrated for each subject.
  Interventions: Biological: CD38 CAR T-cells

INTERVENTIONS:
Biological: CD38 CAR T-cells — Drug: CD38 CAR T-cells Each subject receive CD38 CAR T-cells by intravenous infusion Other Name: CD38 CAR T-cells injection

SUMMARY:
Clinical Study on the Safety and Effectiveness of CD38 CAR-T Cells in the Treatment of CD38-positive Hematological Malignancies

DETAILED DESCRIPTION:
The CAR-T cell injection uses immune cells from healthy donors, and is the final product obtained after CAR genetic modification, cell expansion, culture, screening, preparation, sub-packaging, and release inspection. CD38 is highly expressed in myeloid leukemia, and it has been confirmed that the treatment of targeting CD38 has great potential in the treatment of CD38-positive hematological malignancies. The center intends to apply for a clinical trial of CD38 CAR-T cells to treat CD38-positive hematological malignancies on the basis of preliminary research.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients is histologically diagnosed with CD38-positive AML according to the NCCN Clinical Practice Guidelines in Oncology：Acute Myeloid Leukemia（Version 2.2021）;
* 2. The diagnosis is consistent with r/r CD38 + AML, and includes any of the following conditions:

  1. No CR was obtained after 2 courses of standard chemotherapy
  2. The first induction was CR, but the duration of CR was less than 12 months
  3. No CR was obtained after the first or multiple remedial treatment
  4. Relapse twice or more
* 3. The number of blast cells in bone marrow was more than 5% (morphology) and / or > 1% (flow cytometry);
* 4. No active lung infection, inhaled air oxygen saturation ≥92%;
* 5. The estimated survival time is more than 3 months;
* 6. ECOG score was 0-2;
* 7. The patients or their legal guardians voluntarily participated in the trial and signed the informed consent.

Exclusion Criteria:

* 1. Patients with history of epilepsy or other central nervous system diseases;
* 2. Patients with prolonged QT or severe heart disease;
* 3. Pregnant or lactating women (the safety of this therapy for unborn children is unknown);
* 4. The patients with uncontrolled active infection;
* 5. Active hepatitis B or hepatitis C virus infection;
* 6. Previous application of gene therapy;
* 7. The proiferation rate is less than 5 times response to CD3/CD28 co-stimulation signal;
* 8. Serum creatinine > 2.5mg/dl or ALT / AST > 3 times ULN or bilirubin > 2.0mg/dl;
* 9. Those who suffer from other uncontrolled diseases are not suitable to join the study;
* 10. HIV infection;
* 11. Any situation that the researchers believe may increase the risk of patients or interfere with the test results.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-02-28 (Estimated); Primary Completion 2024-12-05 (Estimated); Study Completion 2024-12-05 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 28 days after CD38 CAR T-cells infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Up to 90 days after CD38 CAR T-cells infusion
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
Concentration of CAR-T cells | From admission to the end of the follow-up, up to 2 years
  In peripheral blood and bone marrow
Disease control rate, DCR | From Day 28 CD38 CAR-T infusion up to 2 years
  The percentage of patients with remission and stable disease after treatment in the total evaluable cases.
Duration of remission, DOR | 24 months post CD38 CAR-T cells infusion
  The time from the first assessment of remission or partial remission of the disease to the first assessment of disease progression or death from any cause
Progression-free survival, PFS | 24 months post CD38 CAR-Tcells infusion
  The time from cell reinfusion to the first assessment of disease progression or death from any cause
Overall survival, OS | From CD38 CAR-T infusion to death，up to 2 years
  The time from the cell reinfusion to death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, PhD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China